CLINICAL TRIAL: NCT06443086
Title: Long-term Survival Outcomes of Duodenal Adenocarcinoma: a Cohort Study With 15-year Single-center Experience
Brief Title: Long-term Outcomes of Duodenal Adenocarcinoma From a Large Cohort
Status: Not yet recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-171
Record Dates: First submitted 2024-05-28; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Gastrointestinal Disease
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Duodenal carcinoma patients: The patients included in this study were drawn from a hospital-based cohort and included cases diagnosed and treated at the facility. Inclusion criteria were histologically confirmed non-ampulla DA, including all stages of disease at diagnosis. Patients were excluded if they had ampulla cancer or other forms of gastrointestinal cancer, had incomplete medical records, or lost follow-up shortly after diagnosis. This rigorous selection process ensured the homogeneity of the study population and the relevance of the findings to non-ampulla DA.
  Interventions: Procedure: Radical operation and perioperative therapy

INTERVENTIONS:
Procedure: Radical operation and perioperative therapy — Surgical intervention, particularly radical excision, was performed for each patient, including the extent of resection and lymph node dissection. Information on adjuvant therapies, such as chemotherapy and radiotherapy, was also recorded, specifying the regimens and durations.

SUMMARY:
The investigators will conducted a hospital-based cohort study in our 15-year experience with DA aimed at investigating the long-term outcomes of the patients with DA, along with analyzing the impact of the tumor characteristics, operations and adjuvant therapy on survival outcomes.

DETAILED DESCRIPTION:
Numerous meta-analyses and systematic reviews have delved into the treatment of DA, yet the majority of the studies retrospective, single-center, and small sample size series, particularly in China. To bridge this knowledge gap, the investigators will conduct a hospital-based cohort study designed to investigate the long-term survival outcomes of the participants with the non-ampulla duodenal adenocarcinoma, and the effects of tumor characteristics, surgery, and adjuvant therapy on survival outcomes.

ELIGIBILITY:
Inclusion criteria:

(1) histologically confirmed non-ampulla DA;

Exclusion criteria:

1. had other gastrointestinal cancer;
2. had incomplete medical records, or lost follow-up shortly after diagnosis;
3. refused clinical data collection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in this study were drawn from a hospital-based cohort and included cases diagnosed and treated at the facility. Inclusion criteria were histologically confirmed non-ampulla DA, including all stages of disease at diagnosis. Patients were excluded if they had ampulla cancer or other forms of gastrointestinal cancer, had incomplete medical records, or lost follow-up shortly after diagnosis. This rigorous selection process ensured the homogeneity of the study population and the relevance of the findings to non-ampulla DA.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Median overall survival time | 2009.10-2023.06
  Median survival is the time it takes half of the individuals in a given study population to reach or exceed a particular end event, calculated from the time an event occurred. Median survival is a statistical index describing the distribution of survival time.
3-year overall survival rate | 2009.10-2023.06
  Three-year survival rate, also known as survival rate, refers to the number of patients with a disease who are still alive at the end of three years of follow-up as a percentage of the number of cases observed
5-year overall survival rate | 2009.10-2023.06
  Five-year survival rate, also known as survival rate, refers to the number of patients with a disease who are still alive at the end of five years of follow-up as a percentage of the number of cases observed

CONTACTS AND LOCATIONS:
Overall Officials: Hao Liu, MD, PhD, Principal Investigator — Department of General Surgery, Nanfang Hospital, Southern Medical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT06443086/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT06443086/ICF_001.pdf